CLINICAL TRIAL: NCT06648083
Title: Analysis of the Factors Influencing the Acquisition of Full Oral Feeding in Very Preterm Infants
Brief Title: Acquisition of Full Oral Feeding and Further Oral Disorders in Extremely Preterm Infants
Acronym: ORAPREM
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2024_002
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Oral Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Food autonomy — Determine the age of acquisition of full oral feeding in extremely premature infants hospitalised in a neonatal unit where that applies a strategy of specific and individualized stimulation of orality.

SUMMARY:
Extremely premature infants (born before 29 weeks) frequently present oral disorders. The management of these patients require assisted ventilation, enteral nutrition, and intensive daily care (procedural pain, exposure to pain, noise, and light), which can have a negative impact on their development. And more specifically on the development of oral skills. In the past decades, the standard of care has evolved and is based on less "aggressive" care and the implication of parents as caregivers. Recent data on the incidence of oral disorders in extremely premature babies are not currently available.

These oral disorders have significant short-term and long-term consequences. During hospitalization, it leads to a delay in the acquisition of full oral feeding, which is defined as the absence of need for tube feeding, and is associated with prolonged hospitalization. It is also associated with a delayed development of orality, which is essential for the proper psychomotor, and cognitive development of premature infants.

Strategies have been proposed to support the acquisition of oral feeding autonomy and to prevent oral feeding disorders, including tactile stimulation of orality consisting in stroking cheeks, peri-oral and intra-oral structures, but there is still no consensus on the best way to support the development of orality in this population.

In this context, a tactile stimulation protocol of orality, has been implemented in the past years, in the neonatal unit of the croix-rousse hospital, based on data published in the literature. It is performed on a daily basis by nurses, and physiotherapists.

In this general context marked by a less aggressive management of orality, and the implementation of an orality stimulation protocol, the main objective of ORAPREM study is to determine the corrected gestational age of oral feeding autonomy in a population of extremely premature infants born recently. Secondary objectives are 1) To analyse risk factors of delay in oral feeding autonomy, to define a subgroup of high-risk infants who could benefit from reinforced interventions to stimulate orality, and 2) To calculate the incidence of oral feeding disorders up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at a gestational age ≤ 28 weeks
* Born between January 1, 2018 and December 31, 2021
* Admitted in the first three days of life in the neonatology department of the Croix-Rousse hospital
* Discharged directly to home (or to a nursery)

Exclusion Criteria:

* Infants re-transferred to another department during hospitalization
* Infants with a severe pathology requiring surgical management in the first weeks of life. Inguinal hernia repair is not concerned
* Severe malformation
* Refusal of the parents

Max Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm newborn born before 28 weeks and hospitalized in the neonatology service of Croix Rousse hospital
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Corrected gestational age at the time of acquisition of full oral feeding | Up to two months
  Corrected gestational age at the time of acquisition of full oral feeding

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Croix Rousse, Lyon, France